CLINICAL TRIAL: NCT06988514
Title: A Single-center, Exploratory, Interventional Clinical Study for Stool Samples Collection in Healthy Participants to Use and Further Advance Some Danone Research Applications
Brief Title: Stool Collection for Model
Acronym: StoColM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24REX0077603
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: A03 - Digestive System; 03 - Bacteria
Keywords: Stool; Microbiota; In vitro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteer collecting stool samples (Experimental): Healthy volunteer collecting and bringing their stool samples to the investigational site.
  Interventions: Other: Standardized stool collection from healthy volunteers

INTERVENTIONS:
Other: Standardized stool collection from healthy volunteers — The only interventions are clinical examination, dietary restrictions and samples collection (stool, and urine for the pregnancy tests (when applicable).

SUMMARY:
Purpose of this study is to collect stool samples from healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged between 18-60 years.
2. 18.5 ≤ BMI < 30 kg/m2.
3. Overtly healthy as determined by the Investigator.
4. Regular bowel movements and a mean stool consistency of 3-5 in Bristol Stool Form Scale (BSFS) during the past week.
5. Able to:

   * Collect their stool samples and delivered at site.
   * Speak and read in French.
   * Comply with the study protocol and to commit to the instructions and restrictions.
   * Refrain from any fermented dairy products throughout the study conduct.
   * Refrain from prebiotic, probiotic or synbiotic supplements during the study.
   * Maintain the dose of other consumed supplements during the study.
   * Limit alcohol consumption to ≤ 2 units (i.e., standard glasses) of alcohol per day with a maximum of 10 units per week during the study.
   * Not change substantially their smoking habits during the study.
6. Written informed consent Form (ICF) signed by the participant.
7. No substantial changes in diet and/or physical activity and/or lifestyle habits, defined as start or stop new foods and/or supplements and/or sports and/or daily habits (i.e., travel, sleeping habits) during the study.
8. Have a personal electronic device compatible and connectable to internet to access the web based MyFood24 site when required.
9. Covered by social security or similar system.
10. Agree to be registered in the National biomedical research file for volunteers.

Exclusion Criteria:

1. Any ongoing metabolic disease, inflammatory disease, hepato-gastrointestinal dis-ease or complications, psychiatric or neurological disorder or other diagnosed by a physician.
2. Any invasive diagnostic and/or therapeutic procedure related to digestion within the past 4 weeks or plan for a digestive surgery during the study, including dental sur-gery, (i.e., from the onset of the wash-out period to the last data collection).
3. General anesthesia during the past 4 weeks or planned during the course of the study.
4. For women in childbearing potential, pregnancy or breastfeeding or plan for preg-nancy during the study.
5. Use of medication that affects the gastrointestinal (GI) function or use of stomach medication within the past 4 weeks or plan to use of any of these during the study.
6. Non-incidental use of > 4 paracetamol tablets (500 mg), nonsteroidal anti-inflammatory drugs (NSAIDs) or aspirin ≤ 2 weeks before the screening visit (V1) or plan of use during the study (if needed, incidental use of ≤ 4 tablets of paracetamol, NSAIDs or aspirin per 2-week period (i.e. ≤ 4 tablets during the refrain period, ≤ 4 tab-lets during the study).
7. Antibiotic, antifungal, antiviral or antiparasitic medication within the past 6 months.
8. Use of any soft drugs, cannabidiol (CBD), plants medicines and/or hard drugs during the study.
9. Participant of another study with investigational or marketed products which could the gut microbiota within the past 4 weeks or plan to participate in such a study dur-ing the study.
10. Participant under guardianship, curatorship, person under judicial protection, family empowerment or future protection mandate.
11. Employees and/or children/family members or relatives of employees of Danone or the participating sites such as medical, pharmacy, dental and nursing students, sub-ordinate hospital and laboratory personnel, employees of the Investigator or of the Sponsor, members of the armed forces, and persons kept in detention.
12. Having received, during the last 12 months, indemnities for participation into clinical study exceeding the annual threshold of 6000€ (including participation to this study).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2025-06-19 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Collect enough acceptable stool samples | After 14 days of refrain period

OTHER OUTCOMES:
The objective of this study is to collect enough acceptable stool samples from healthy participants to develop the three Danone research applications. | After 14 days of refrain period
  So, the main outcome parameter of this study is the number of acceptable samples for further studies:
  n= 50 samples for the in vitro colonic gas model. n= 72 samples for Danone's sequencing platform. n= 72 samples for Danone's strain collection.
Dietary intakes of the previous day of the faecal samples collection for V2 (collected using my Food24 after sample delivery) and V3 (if applicable). | After 14 days of refrain period

CONTACTS AND LOCATIONS:
Locations (1):
- CEN Experimental, Dijon, France

IPD SHARING:
Plan to Share IPD: No